CLINICAL TRIAL: NCT07059728
Title: Uso de Lentillas de Alto Flujo en Procedimientos de sustitución de válvula aórtica transcatéter. Impacto en Las Complicaciones Respiratorias y Biomarcado- Res y Resultados clínicos. TAVR-Highflow
Brief Title: High Flow Nasal Oxygenation in Transcatheter Aortic Valve Replacement Procedures. TAVR-Highflow II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2025/0514
Record Dates: First submitted 2025-06-18; First posted 2025-07-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-06

CONDITIONS: Aortic Stenosis Treated With TAVI; Sedation; Aged; Hemodynamics
Keywords: Aortic Stenosis; TAVR; Sedation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HFNO group (Experimental): Patients recieving high flow nasal oxygenation
  Interventions: Device: Oxygen therapy during sedation provided via high nasal cannulae (60L/min at 60% FiO2)
- Control group (Active Comparator): Patients recieving standard of care oxygen theraphy (5L/min via nasal cannulae)
  Interventions: Device: Oxygen therapy during sedation delivered via nasal cannulae at 5L/min

INTERVENTIONS:
Device: Oxygen therapy during sedation provided via high nasal cannulae (60L/min at 60% FiO2) — Intervention group: Oxygen therapy during sedation provided via high nasal cannulae (60L/min at 60% FiO2)
  Arms: HFNO group
Device: Oxygen therapy during sedation delivered via nasal cannulae at 5L/min — Control group: Oxygen therapy during sedation delivered via nasal cannulae at 5L/min
  Arms: Control group

SUMMARY:
Transcatheter aortic valve replacement (TAVR) has revolutionized the treatment of patients with aortic valve disease. TAVR is a less invasive treatment compared to the conventional surgical approach through median sternotomy.

Patients selected for this procedure often have a profile associated with multiple comorbidities which predispose them to certain complications.

TAVI procedures were initially performed under general anesthesia. However, due to improved procedure times and anesthetic techniques, sedation has become the current trend to preform them.

When sedation for these procedures requires deep planes, hypoxia is more likely to occur due to respiratory depression, apnea, or airway obstruction. This is even more common in TAVR patients population, as obesity, sleep apnea, elevated ASA classification, advanced age, and combined cardiorespiratory disease are highly prevalent.

For all these reasons, TAVR constitutes a risky procedure, presenting a profile of patients undergoing this procedure that can also be considered high risk.

The provision of supplemental oxygen through nasal cannulae or face masks can prevent the development of hypoxia. Unfortunately, non-humidified nasal oxygen cannot exceed 2-5 L/min without causing damage to the nasal mucosa, and the percentage of oxygen delivered through variable-flow face masks is unpredictable.

On the other hand, high-flow nasal oxygen therapy (HFNO) can provide humidified gas flow rates of up to 70 L/min through specially adapted nasal cannulae and reliably deliver oxygen concentrations between 21% and 100%. The use of HFNC could be justified in this context and could improve the outcomes and safety of these procedures, increasing oxygen content and minimizing hypercapnia.

The study's hypothesis is HFNO will prevent hypoxemia and control hypercapnia during sedation for transcatheter aortic valve implantation (TAVI) better than conventional oxygen theraphy. Clinical and serological biomarkers of tissue injury will decrease with the use of HFNO. Clinical complications will decrease with the use of HFNO.

The study population would be all patients >18 years of age undergoing TAVI procedure and who agree to participate in the study in 8 centers in Barcelona.

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVR) has revolutionized the treatment of patients with aortic valve disease. TAVR is a less invasive treatment compared to the conventional surgical approach through median sternotomy. These technological advances have enabled a minimally invasive anesthetic approach that avoids mechanical ventilation, central line insertion, and urinary catheterization in most patients undergoing TAVR.

However, patients selected for this procedure often have a profile associated with multiple comorbidities such as pulmonary disease, ischemic coronary artery disease, and atherosclerosis of the carotid and renal arteries, which predispose them to certain complications.

Acute kidney injury (4%-35%), ischemic stroke (1%-3%), acute heart failure (7%-24%), and hypoxemia with hypercapnia are the most common perioperative complications. The overall 30-day mortality rate is 2.2%.

Because they are considered high-risk (both due to the procedure and the type of patient undergoing this procedure) and due to their duration, TAVI procedures were initially performed under general anesthesia. With improved procedure times and improved anesthetic techniques, the trend is to attempt to perform these procedures under deep sedation. As in many settings, sedation for diagnostic and/or therapeutic procedures can be achieved with a variety of medications, the goal of which is sedation to enable procedural success. The development and advancement of procedures as an alternative to surgery and/or more invasive diagnostic and therapeutic procedures means that the use of less invasive techniques is becoming increasingly common. Depending on the procedure, sedation may be required. However, despite the less invasive nature of these tests, deep sedation is frequently required for these procedures.

Deep sedation techniques have developed alongside technological advances that enable the provision of complex diagnostic and therapeutic procedures, often performed in settings outside the operating room. These settings include procedure rooms, radiology departments, outpatient departments, emergency rooms, surgical facilities, interventional cardiology departments, and so on. Deep sedation is used to support and enable the performance of these procedures. Enthusiasm for providing sedation for these procedures in a non-OR setting was tempered by an increase in mortality in non-OR areas, even leading one author to describe this as the "Wild West" of surgical and anesthetic practice. This required both professionals and regulatory authorities have developed increased oversight to improve the quality of care for out-of-the-operative procedures.

When sedation for these procedures requires deep planes, hypoxia is more likely to occur due to respiratory depression, apnea, or airway obstruction. This is even more common in patients at risk due to obesity, sleep apnea, elevated ASA classification, age >60 years, and combined cardiorespiratory disease. The reported incidence of hypoxia ranges from 10% to 70%, depending on the definition of hypoxia used. The risk of hypoxia further increases with the duration of the procedure.

The risk of periprocedural hypoxia can be reduced by monitoring respiratory and sedation parameters. However, even the most effective monitoring and standards of care may not be sufficient to reverse the respiratory compromise caused by deep sedation. Deep sedation affects the respiratory system through effects on normal cardiorespiratory physiology. These changes include a drop in respiratory rate, tidal volume, and changes in cardiorespiratory dynamics, and these effects are further affected by patient positioning. Subjects with cardiorespiratory diseases, such as pulmonary hypertension and chronic respiratory diseases, are particularly at risk for a critical decline in function.

The provision of supplemental oxygen through nasal cannulae or face masks can prevent the development of hypoxia. Unfortunately, non-humidified nasal oxygen cannot exceed 2-5 L/min without causing damage to the nasal mucosa, and the percentage of oxygen delivered through variable-flow face masks is unpredictable.

High-flow nasal oxygen therapy (HFNO), which is also unique in that it is humidified, was developed to provide flow rates of up to 70 L/min through specially adapted nasal cannulae and reliably delivers oxygen concentrations between 21% and 100%. Many operators are finding that combining deep planes of sedation with HFNC reduces the risk of periprocedural hypoxia. HFNC reduces the work of breathing, physiological dead space and provides an element of positive end-expiratory airway pressure.

HFNO has the potential to reduce procedural hypoxic events, procedural interruptions, and increase therapeutic success. However, although not all trials have concluded that HFNO improves safety compared to standard nasal oxygen therapy, the experience of most operators is positive.

The additional cost of HFNO may be a limiting factor for its use during procedural sedation, but it may be justified in high-risk procedures and patients with risk factors (already discussed), as it improves safety and quality of care. Deep sedation now allows complex diagnostic and therapeutic procedures to be performed outside the operating room in high-risk patients, but it is not without risk, and tools must be developed to mitigate the possibility of such risk.

For all the reasons stated above, TAVI constitutes a risky procedure, presenting a profile of patients undergoing this procedure that can also be considered high risk. The use of HFNC could be justified in this context and could improve the outcomes and safety of these procedures.

The use of HFNC during sedation for TAVI could increase oxygen content and minimize hypercapnia, which frequently occur. This may have two potential benefits: one in terms of facilitating patient tolerance to anesthetic sedation; and the other in optimizing oxygen delivery to organs such as the brain, kidneys, and myocardium. Currently, the profile of patients typically proposed for TAVI is those with aortic disease and significant morbidity and/or older age, who have been ruled out for conventional surgery. These patients are more likely to develop periprocedural complications, being specially sensitive to them.

In a recent study conducted in the United Kingdom, the use of HFNO with a FiO2 of 30% was associated with an 18% reduction in desaturation episodes; however, a decrease in hypoxemia measured by arterial oxygen levels could not be observed.

In a recent randomized clinical trial conducted at the Hospital Clínic in Barcelona (currently under review), the use of HFNO with a FiO2 of 60% was associated with a 31% reduction in desaturation episodes, higher arterial oxygen levels, and improved postoperative renal function, both analytically (measured by creatinine and glomerular filtration rate) and clinically (a 10% reduction in the incidence of renal failure according to VARC criteria).

However, several questions remain to be determined. First, a potential impact (both clinical and analytical) on preventing damage to other target organs (brain and heart). Second, the identification of patient subgroups at higher risk of desaturation and hypoxemia during deep sedation and who, consequently, may benefit more from HFNC treatment. Finally, there is still no data to assess the clinical impact of HFNC on clinical variables such as mortality, hospital stay, and reduction of postoperative complications (stroke, delirium, heart failure, etc.).

The justification for the study would be the use of HFNC, a therapy already available in healthcare centers but not widely used for these procedures. The risks of its use are comparable to those of conventional nasal oxygen therapy. Potential benefits would include a reduction in respiratory complications, a potential improvement in organ-specific biomarker levels, and a potential reduction in clinical cardiological, neurological, and renal complications, as well as an improvement in hospital stay and periprocedural mortality.

The study population would be all patients >18 years of age undergoing TAVI procedure and who agree to participate in the study in 8 centers in Barcelona.

ELIGIBILITY:
Inclusion Criteria:

* Transfemoral TAVR elective procedure
* Age >18 years

Exclusion Criteria:

* Patients under 18 years of age
* Refusal to participate
* Known allergy to propofol or remifentanil.
* Non-femoral surgical access.
* Presence of a basal skull fracture or pneumothorax
* Procedure duration < 45 minutes
* Previously planned general anaesthesia approach due to patient's condition or procedural technical reasons
* Need to convert to general anesthesia for non-respiratory complications within 45 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | From enrollment to 30 days after intervention
  Reduction in complications at 30 days post-procedure). Classic composite variable that includes: 30-day post-procedure mortality, need for hospital readmission due to acute heart failure, incidence of stroke, and incidence of acute kidney injury.
Win ratio | From enrollment to 30 days after the intervention ends
  Win ratio analysis for outcomes: 30-day post-procedure mortality, need for hospital readmission for acute heart failure, incidence of acute stroke, incidence of acute kidney injury, and quality of life (measured by the Kansas Questionnaire)

SECONDARY OUTCOMES:
Number of Desaturation episodes | From enrollment until end of TAVR procedure
  Pulse oximetry values inferior to 93% for a period of more than 10 seconds.
Desaturation incidence | From enrollment until the end of TAVR procedure
  Probability of presenting at least 1 episode of desaturation
PaO2 | At enrollment and at 45 minutes after enrollment
  Arterial partial pressure oxygen
PaCO2 | At enrollment and at 45 minutes after enrollment.
  CO2 arterial partial pressure
Neuronal Specific Enolase | At enrollment and at 8 hours after enrollment.
  Serological Neuronal Specific Enolase levels.
Creatinine | At enrollment and at 8 hours after enrollment.
  Creatinine serological levels
Troponin | At enrollment and at 8 hours after enrollment.
  Ultra-sensitive Troponin serological levels
NT-proBNP | At enrollment and at 8 hours after enrollment.
  NT-proBNP serological levels
Number of patients presenting with respiratory depression | From enrollment until the end of TAVR procedure
  Any desaturation episode that leads to patient's manual ventilation from responsible anesthesiologyst in order to mantain patients well being.
Vasopressors | From enrollment until the end of TAVR procedure.
  Drugs used to mantain mean blood pressure levels above 65mmHg. Drug used and dose administered.
Propofol and remifentanil | From enrollment until the end of TAVR procedure
  Drugs used to induce and mantain hypnosis. Total amount of propofol and remifentanil administered during the procedure
Procedural duration | Procedure (Time from start of sedation to when sedation drugs are stopped)
  Time of duration of sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Scheuermann S, Tan A, Govender P, Mckie M, Pack J, Martinez G, Falter F, George S, A Klein A. High-flow nasal oxygen vs. standard oxygen therapy for patients undergoing transcatheter aortic valve replacement with conscious sedation: a randomised controlled trial. Perioper Med (Lond). 2023 Apr 14;12(1):11. doi: 10.1186/s13741-023-00300-8. PMID 37060038
- [Background] Turnbull D. High-flow nasal oxygen, procedural sedation, and clinical governance. Minerva Anestesiol. 2022 May;88(5):407-410. doi: 10.23736/S0375-9393.21.16078-X. Epub 2021 Sep 16. PMID 34527411
- [Background] Riddell Z, Pressler N, Siau K, Mulder CJJ, Shalmani HM, Downs A, Gait A, Ishaq S. Feasibility of high-flow nasal oxygen therapy and two-stage sedation during endoscopic hypopharyngeal therapy. JGH Open. 2020 May 16;4(4):743-748. doi: 10.1002/jgh3.12348. eCollection 2020 Aug. PMID 32782965
- [Background] Riccio CA, Sarmiento S, Minhajuddin A, Nasir D, Fox AA. High-flow versus standard nasal cannula in morbidly obese patients during colonoscopy: A prospective, randomized clinical trial. J Clin Anesth. 2019 May;54:19-24. doi: 10.1016/j.jclinane.2018.10.026. Epub 2018 Nov 2. PMID 30391445
- [Background] Kim SH, Bang S, Lee KY, Park SW, Park JY, Lee HS, Oh H, Oh YJ. Comparison of high flow nasal oxygen and conventional nasal cannula during gastrointestinal endoscopic sedation in the prone position: a randomized trial. Can J Anaesth. 2021 Apr;68(4):460-466. doi: 10.1007/s12630-020-01883-2. Epub 2021 Jan 6. PMID 33403549
- [Background] Sago T, Harano N, Chogyoji Y, Nunomaki M, Shiiba S, Watanabe S. A nasal high-flow system prevents hypoxia in dental patients under intravenous sedation. J Oral Maxillofac Surg. 2015 Jun;73(6):1058-64. doi: 10.1016/j.joms.2014.12.020. Epub 2014 Dec 30. PMID 25799356
- [Background] Lin Y, Zhang X, Li L, Wei M, Zhao B, Wang X, Pan Z, Tian J, Yu W, Su D. High-flow nasal cannula oxygen therapy and hypoxia during gastroscopy with propofol sedation: a randomized multicenter clinical trial. Gastrointest Endosc. 2019 Oct;90(4):591-601. doi: 10.1016/j.gie.2019.06.033. Epub 2019 Jul 3. PMID 31278907
- [Background] Teng WN, Ting CK, Wang YT, Hou MC, Chang WK, Tsou MY, Chiang H, Lin CL. High-Flow Nasal Cannula and Mandibular Advancement Bite Block Decrease Hypoxic Events during Sedative Esophagogastroduodenoscopy: A Randomized Clinical Trial. Biomed Res Int. 2019 Jul 16;2019:4206795. doi: 10.1155/2019/4206795. eCollection 2019. PMID 31380421
- [Background] Ischaki E, Pantazopoulos I, Zakynthinos S. Nasal high flow therapy: a novel treatment rather than a more expensive oxygen device. Eur Respir Rev. 2017 Aug 9;26(145):170028. doi: 10.1183/16000617.0028-2017. Print 2017 Sep 30. PMID 28794144
- [Background] Wen Z, Wang W, Zhang H, Wu C, Ding J, Shen M. Is humidified better than non-humidified low-flow oxygen therapy? A systematic review and meta-analysis. J Adv Nurs. 2017 Nov;73(11):2522-2533. doi: 10.1111/jan.13323. Epub 2017 May 30. PMID 28440960
- [Background] Wagstaff TA, Soni N. Performance of six types of oxygen delivery devices at varying respiratory rates. Anaesthesia. 2007 May;62(5):492-503. doi: 10.1111/j.1365-2044.2007.05026.x. PMID 17448063
- [Background] Raman V, Raman V, Tobias JD. Dexmedetomidine and Pulmonary Hype- rtension: A Case Report and Review of the Literature. J Med Cases. 2013;4(7):481-484. doi:10.4021/jmc.v4i7.1279
- [Background] Wang CY, Ling LC, Cardosa MS, Wong AK, Wong NW. Hypoxia during upper gastrointestinal endoscopy with and without sedation and the effect of pre-oxygenation on oxygen saturation. Anaesthesia. 2000 Jul;55(7):654-8. doi: 10.1046/j.1365-2044.2000.01520.x. PMID 10919420
- [Background] Bell JK, Laasch HU, Wilbraham L, England RE, Morris JA, Martin DF. Bispectral index monitoring for conscious sedation in intervention: better, safer, faster. Clin Radiol. 2004 Dec;59(12):1106-13. doi: 10.1016/j.crad.2004.04.008. PMID 15556593
- [Background] Saunders R, Struys MMRF, Pollock RF, Mestek M, Lightdale JR. Patient safety during procedural sedation using capnography monitoring: a systematic review and meta-analysis. BMJ Open. 2017 Jun 30;7(6):e013402. doi: 10.1136/bmjopen-2016-013402. PMID 28667196
- [Background] Qadeer MA, Rocio Lopez A, Dumot JA, Vargo JJ. Risk factors for hypoxemia during ambulatory gastrointestinal endoscopy in ASA I-II patients. Dig Dis Sci. 2009 May;54(5):1035-40. doi: 10.1007/s10620-008-0452-2. Epub 2008 Nov 12. PMID 19003534
- [Background] van Schaik EPC, Blankman P, Van Klei WA, Knape HJTA, Vaessen PHHB, Braithwaite SA, van Wolfswinkel L, Schellekens WM. Hypoxemia during procedural sedation in adult patients: a retrospective observational study. Can J Anaesth. 2021 Sep;68(9):1349-1357. doi: 10.1007/s12630-021-01992-6. Epub 2021 Apr 20. PMID 33880728
- [Background] Wax D. Regulatory issues in office-based surgery and anesthesia. Semi- nars in Anesthesia, Perioperative Medicine and Pain. 2006;25(1):25-31. doi:10.1053/J.SANE.2005.11.005
- [Background] Quattrone MS. Is the physician office the wild, wild west of health care? J Ambul Care Manage. 2000 Apr;23(2):64-73. doi: 10.1097/00004479-200004000-00009. PMID 10848394
- [Background] Puijk RS, Ziedses des Plantes V, Nieuwenhuizen S, Ruarus AH, Vroomen LGPH, de Jong MC, Geboers B, Hoedemaker-Boon CJ, Thone-Passchier DH, Gercek CC, de Vries JJJ, van den Tol PMP, Scheffer HJ, Meijerink MR. Propofol Compared to Midazolam Sedation and to General Anesthesia for Percutaneous Microwave Ablation in Patients with Hepatic Malignancies: A Single-Center Comparative Analysis of Three Historical Cohorts. Cardiovasc Intervent Radiol. 2019 Nov;42(11):1597-1608. doi: 10.1007/s00270-019-02273-y. Epub 2019 Jun 26. PMID 31243542
- [Background] Horn P, Hellhammer K, Minier M, Stenzel MA, Veulemans V, Rassaf T, Luedike P, Pohl J, Balzer J, Zeus T, Kelm M, Westenfeld R. Deep sedation Vs. general anesthesia in 232 patients undergoing percutaneous mitral valve repair using the MitraClip(R) system. Catheter Cardiovasc Interv. 2017 Dec 1;90(7):1212-1219. doi: 10.1002/ccd.26884. Epub 2017 Jan 23. PMID 28112459
- [Background] Raffay V, Fišer Z, Samara E, et al. Challenges in procedural sedation and anal- gesia in the emergency department. Journal of Emergency and Critical Care Medicine. 2020;8:27-27. doi:10.21037/jeccm-19-212
- [Background] Cote GA, Hovis RM, Ansstas MA, Waldbaum L, Azar RR, Early DS, Edmundowicz SA, Mullady DK, Jonnalagadda SS. Incidence of sedation-related complications with propofol use during advanced endoscopic procedures. Clin Gastroenterol Hepatol. 2010 Feb;8(2):137-42. doi: 10.1016/j.cgh.2009.07.008. Epub 2009 Jul 14. PMID 19607937
- [Background] Anwaruddin S, Desai ND, Vemulapalli S, Marquis-Gravel G, Li Z, Kosinski A, Reardon MJ. Evaluating Out-of-Hospital 30-Day Mortality After Transfemoral Transcatheter Aortic Valve Replacement: An STS/ACC TVT Analysis. JACC Cardiovasc Interv. 2021 Feb 8;14(3):261-274. doi: 10.1016/j.jcin.2020.10.027. PMID 33541537
- [Background] Jakulla RS, Gunta SP, Huded CP. Heart Failure after Aortic Valve Replacement: Incidence, Risk Factors, and Implications. J Clin Med. 2023 Sep 19;12(18):6048. doi: 10.3390/jcm12186048. PMID 37762989
- [Background] Shekhar S, Isogai T, Agrawal A, Kaw R, Mahalwar G, Krishnaswamy A, Puri R, Reed G, Mentias A, Kapadia S. Outcomes and Predictors of Stroke After Transcatheter Aortic Valve Replacement in the Cerebral Protection Device Era. J Am Heart Assoc. 2024 Aug 6;13(15):e034298. doi: 10.1161/JAHA.124.034298. Epub 2024 Aug 5. PMID 39101495
- [Background] Zaleska-Kociecka M, Dabrowski M, Stepinska J. Acute kidney injury after transcatheter aortic valve replacement in the elderly: outcomes and risk management. Clin Interv Aging. 2019 Jan 21;14:195-201. doi: 10.2147/CIA.S149916. eCollection 2019. PMID 30718946